CLINICAL TRIAL: NCT05684601
Title: Analysis Impact of 3D Intraoral Scanning on Postsurgical Evaluation of Mandibular Third Molar Surgery Using Piezosurgery Versus Traditional Rotating Instrumentations
Brief Title: Impact of 3D Intraoral Scanning on Postsurgical Evaluation of Mandibular Third Molar Surgery
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Catania (Other)
Responsible Party: Principal Investigator, Gaetano Isola, Researcher, University of Catania
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 65-22-PO
Record Dates: First submitted 2022-12-26; First posted 2023-01-13 (Actual); Last update posted 2023-01-13 (Actual); Status verified 2023-01

CONDITIONS: Third Molar Surgery; Impacted Third Molar Tooth

STUDY DESIGN:
Intervention Model Description: Thee primary outcome was postoperative pain, evaluated using the visual analogue scale (VAS) score at Baseline, 1, 2, 5, 7, 10, 14 and 28 days following surgery in subject treated for third molar surgery with piezoelectric surgery or rotating drills. The secondary outcomes chosen were changes in postoperative swelling and maximum mouth opening values compared to preoperative ones.
Who Masked: Participant, Care Provider
Masking Description: Treatment performed with sealed envelopes
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- rotating drills device (Placebo Comparator): Third molar surgery performed with traditional rotating devices
  Interventions: Device: Third molar surgery
- Piezoelectric device (Active Comparator): Third molar surgery performed with piezoelectric surgery device
  Interventions: Device: Third molar surgery

INTERVENTIONS:
Device: Third molar surgery — It was extracted one impacted mandibular third molar per patient with piezoelectric or rotating drills device

SUMMARY:
The aim of this study was to analyze the effectiveness of piezoelectric surgery and traditional rotating device in reducing perioperative sequelae after impacted mandibular third molar surgery in 56 subjects. Ni All subjects were randomly allocated to receive one treatment.

DETAILED DESCRIPTION:
The aim of this study was to analyze the effectiveness of piezoelectric surgery and traditional rotating device in reducing perioperative sequelae after impacted mandibular third molar surgery. Fifty-six patients who needed surgical extraction of an impacted mandibular third molar were selected for the study. All subjects were randomly allocated to receive one of the following surgical treatments piezoelectric surgery (n = 28), traditional surgery with rotating device (n = 28). The primary outcome was postoperative pain, evaluated using the visual analogue scale (VAS) score at baseline, 1, 2, 5, 7, 10 and 14 and 28 days following surgery. The secondary outcomes chosen were changes in postoperative swelling and maximum mouth opening values compared to preoperative ones.

ELIGIBILITY:
Inclusion Criteria:

* aged between 18 and 32 years;
* good general health;
* the presence of one impacted third molar in the mandible with a class II position, type B impaction;
* absence of pericoronitis or signs of inflammation during the last 30 days. Panoramic radiographs were used to determine tooth position.

Exclusion Criteria:

* the presence of any systemic disease;
* consumption of oral contraceptives or other medications;
* consumption of any immunosuppressive or anti-inflammatory drugs during the 3 months prior to the study;
* status of pregnancy or lactation;
* previous history of excessive drinking;
* allergy to local anesthetic;
* smoking habit.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 56 (Actual)
Dates: Start 2020-09-15 (Actual); Primary Completion 2022-10-20 (Actual); Study Completion 2022-10-20 (Actual)

PRIMARY OUTCOMES:
Visual analogue Scale (VAS), values 1-10 | 1- and 3-months
  Evaluation of VAS value changes at baseline and follow-up session

CONTACTS AND LOCATIONS:
Overall Officials: Gaetano Isola, Principal Investigator — University of Catania
Locations (1):
- AOU Policlinico G. Rodolico, Catania, Italy

IPD SHARING:
Plan to Share IPD: Yes
Study protocol
Supporting Information: Study Protocol
Time Frame: 1-year
Access Criteria: Publication on pubmed